CLINICAL TRIAL: NCT05506449
Title: Early Impella® Support in Patients With ST-Segment Elevation Myocardial Infarction Complicated by Cardiogenic Shock: The RECOVER IV Trial
Brief Title: The RECOVER IV Trial
Acronym: RECOVER IV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Given the findings from the DanGer Shock RCT, the RECOVER IV independent DSMB believes that equipoise for randomization in the RECOVER IV Trial no longer exists and has recommended that the RECOVER IV Trial be permanently discontinued.
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABMD-CIP-22-02
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI); Cardiogenic Shock
Keywords: Cardiovascular Diseases; Myocardial Infarction; Heart Failure; Exception From Informed Consent (EFIC); Cardiogenic Shock
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Shock, Cardiogenic; Cardiovascular Diseases; Myocardial Infarction; Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized, controlled, open-label two-arm trial with an adaptive design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Arm (Active Comparator): Subjects randomized to the Control Arm will be treated based on recommendations for cardiogenic shock in the contemporary AHA/ACC/SCAI and ESC Practice Guidelines for STEMI and Heart Failure Management and local standard of care.
  Interventions: Other: Standard of Care
- Treatment Arm (Experimental): Subjects randomized to the Treatment Arm will receive hemodynamic support using an Impella-based treatment strategy initiated prior to percutaneous coronary intervention (PCI).
  Interventions: Device: Impella CP®

INTERVENTIONS:
Device: Impella CP® — Subjects randomized to the Treatment Arm will undergo Impella CP placement prior to PCI. Right heart catheterization will be performed prior to or immediately after PCI.
  Use of IABP will not be allowed in the Treatment Arm.
  Arms: Treatment Arm
Other: Standard of Care — This may include inotropes and/or vasopressors. An IABP may or may not be used according to local practice and the specific condition of each individual patient. If an IABP is used, it may be placed prior to or after PCI, and its timing of explant is left to the discretion of the Investigator.
  Arms: Control Arm

SUMMARY:
The purpose of this study is to assess whether hemodynamic support with an Impella-based treatment strategy initiated prior to percutaneous coronary intervention (PCI) in patients with ST-Segment Elevation Myocardial Infarction (STEMI)-Cardiogenic Shock (CS) improves survival and functional outcomes compared to a non-Impella-based treatment strategy.

DETAILED DESCRIPTION:
To demonstrate that hemodynamic support with an Impella-based treatment strategy initiated prior to PCI, when compared with a non-Impella-based standard of care treatment strategy reduces all-cause mortality at 30 days in patients with STEMI-CS.

ELIGIBILITY:
Inclusion Criteria:

1. Cardiogenic shock with onset ≤12 hours after STEMI and prior to index PCI, as defined by having both the following:

   1. Persistent SBP <90 mmHg for ≥30 minutes despite fluid resuscitation or pressors/inotropes required to maintain SBP ≥90 mmHg and
   2. Signs of impaired organ perfusion (cool extremities and/or altered mental status)
2. One of the following must be present on a standard 12-lead electrocardiogram (ECG):

   1. ST-segment elevation (≥2 mm elevation of ST-segments in ≥2 contiguous leads without left bundle branch block) or
   2. Anterior (V1-V4) ST-segment depression ≥2 mm in ≥2 contiguous leads consistent with a possible posterior infarction AND coronary angiogram prior to randomization showing acute total or subtotal occlusion of the proximal circumflex artery or
   3. aVR ST-segment elevation ≥2 mm without anterior ST-segment elevation AND coronary angiogram prior to randomization confirming left main culprit lesion

      * NOTE: Patients with isolated RV infarction are excluded from this Protocol. If a patient qualifies with cardiogenic shock with only inferior ST-segment elevation, pre-randomization assessment of LV function must be obtained with either point of care echocardiography or contrast left ventriculography to demonstrate a LVEF ≤40% for the patient to be eligible for randomization.
3. Intended emergent PCI to treat the STEMI
4. Subject is able to and agrees to provide written informed consent. If the subject is unable to be consented because of their extreme illness and a legally authorized representative (LAR) is present, the LAR must agree and provide written informed consent. If the subject is unable to provide consent because of their extreme illness and an LAR is not present, the patient may be randomized under Exception from Informed Consent (EFIC) Guidance

Exclusion Criteria:

1. High suspicion for isolated right ventricular infarct confirmed with ECG lead V4R
2. Cardiogenic shock with either of the following:

   1. High-grade atrioventricular block (heart rate (HR) <50 bpm)

      * NOTE: If patient is paced, via temporary or permanent pacemaker, and still in shock, they are still eligible
   2. Isolated narrow complex supraventricular tachycardia with ventricular response >170 bpm or ventricular tachyarrhythmia with ventricular response >150 bpm
3. Known mechanical complications of acute myocardial infarction (AMI) that may cause cardiogenic shock such as free wall rupture, cardiac tamponade, ventricular septal defect or papillary muscle rupture with acute mitral regurgitation
4. Left ventricular function (LVEF >40%) on echocardiography or LV-gram (if performed) indicating shock due to another cause (e.g., RV infarction as the principal cause of shock, hypovolemia, sepsis or high cardiac output shock)
5. Severe bilateral peripheral arterial disease precluding femoral Impella CP insertion (femoral angiogram required) NOTE: Impella insertion via a non-femoral arterial route is not permitted in this Protocol.
6. IABP, Impella or other mechanical circulatory support already in place for present indication (pre-randomization)
7. Known end-stage renal disease, receiving dialysis
8. Severe aortic stenosis, or moderate or worse aortic regurgitation or prior self-expanding transcatheter aortic valve replacement (TAVR), or surgically placed mechanical valve, if known
9. Acute or chronic aortic dissection, if known
10. Large or mobile LV thrombus, if known
11. Prior PCI for the present infarction
12. Prior PCI or coronary artery bypass graft (CABG) within 1 year, if known
13. Ongoing cardiopulmonary resuscitation (CPR)
14. Not obeying verbal commands after preadmission or in-hospital cardiac arrest

    * NOTE: (i) A positive and appropriate response to commands must be repeatable on at least two (2) instances to rule out reflex response to voice (ii) Intubated subjects may be enrolled if:

      1. They did not have a cardiac arrest and were following verbal commands prior to intubation or
      2. They are clearly following verbal commands after intubation
15. Prior stroke with permanent, significant neurological defect
16. Prior intracranial hemorrhage or known intracerebral mass, aneurysm or fistula
17. Acute or suspected stroke prior to randomization
18. Active infection requiring oral or intravenous antibiotics
19. Prior heparin-induced thrombocytopenia, if known
20. Other severe, concomitant disease with limited life expectancy <1 year (other than cardiogenic shock)
21. Pregnancy, known or suspected
22. Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device that has not reached its primary endpoint or any cardiogenic shock trial other than a registry
23. If known, subject has previously been symptomatic with or hospitalized for COVID-19 unless he/she has been discharged (if hospitalized) and asymptomatic for ≥4 weeks and has returned to his/her prior baseline (pre-COVID) clinical condition
24. Subject has other medical, social or psychological conditions that, in the opinion of the Investigator, compromises the subject's ability to comply with study procedures (e.g., dementia, severe alcohol or substance abuse)
25. Patient belongs to a vulnerable population [Vulnerable patient populations may include individuals with mental disability, persons in nursing homes, impoverished persons, homeless persons, nomads, refugees and those permanently incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces and persons kept in detention]
26. Patient is wearing a bracelet or other item indicating their wishes to decline participation in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-10-28 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality | 30 Days

SECONDARY OUTCOMES:
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 30 Days
Days Alive Out-of-Hospital | 6 Months
Mean Change in Health-Related Quality of Life, as measured by Kansas City Cardiomyopathy Questionnaire | 1 Year

OTHER OUTCOMES:
All-Cause Mortality | At hemodynamic stability and when the subject is no longer hospitalized, 6 Months, 1 Year
MACCE | At hemodynamic stability when the subject is no longer hospitalized, 6 Months, 1 Year
Days Alive Out-of-Hospital | 30 Days, 6 Months
Mean Change in Health-Related Quality of Life, as measured by Kansas City Cardiomyopathy Questionnaire | 30 Days Post-Discharge, 6 Months
Mean Change in Health-Related Quality of Life, as measured by Rose Dyspnea Score | 30 Days Post-Discharge, 6 Months, 1 Year
Mean Change in Health-Related Quality of Life, as measured by EQ-5D-5L | 30 Days Post-Discharge, 6 Months, 1 Year
Left Ventricular Ejection Fraction (LVEF) | 30 Days, 6 Months
Estimated Glomerular Filtration Rate (eGFR) | At hemodynamic stability when the subject is no longer hospitalized, 30 Days, 6 Months, 1 Year
Number of Participants with need for In-Hospital Hemodialysis or Continuous Renal Replacement Therapy (CRRT) | At hemodynamic stability when the subject is no longer hospitalized
Number of Participants with need for Dialysis Post-Index Hospitalization | 30 Days, 6 Months, 1 Year
Number of Participants with any Dialysis | 30 Days, 6 Months, 1 Year
All-Cause Hospitalizations | 30 Days, 6 Months, 1 Year
Cardiovascular Hospitalizations | 30 Days, 6 Months, 1 Year
Heart Failure Hospitalizations | 30 Days, 6 Months, 1 Year
Number of Participants with new Implantable Cardioverter Defibrillator (ICD) or Cardiac Resynchronization Therapy (CRT) Implant | At hemodynamic stability when the subject is no longer hospitalized, 30 Days, 6 Months, 1 Year
Number of Participants with Left Ventricular Assist Device (LVAD) or Heart Transplant (including United Network for Organ Sharing (UNOS) 1/2 listing) | At hemodynamic stability when the subject is no longer hospitalized, 30 Days, 6 Months, 1 Year
Repeat Target Vessel Revascularization (TVR) | 30 Days, 6 Months, 1 Year
Acute Kidney Injury (AKI) | within 7 Days Post-Percutaneous Coronary Intervention (PCI)
Disability Assessed using the Modified Rankin Scale | At hemodynamic stability when the subject is no longer hospitalized, 30 Days, 6 Months, 1 Year
30-day survival with mRS score ≤3 | 30 day
Number of Participants with Neurologic Academic Research Consortium (NeuroARC) Type 1 Stroke | At hemodynamic stability when the subject is no longer hospitalized
Major Bleeding | Shock Academic Research Consortium (SHARC) Types 3-5, At hemodynamic stability when the subject is no longer hospitalized
Major Vascular Complications | SHARC Definition, At hemodynamic stability when the subject is no longer hospitalized
Major Hemolysis | At hemodynamic stability when the subject is no longer hospitalized
Major Cath Lab Complications | All adverse events will be recorded and documented through 1 year follow up or study completion
  Intubation; new bradyarrhythmia requiring a temporary pacemaker; ventricular arrhythmias requiring cardioversion or defibrillation; persistent severe hypotension or heart failure requiring escalation beyond the randomized study devices (Impella CP in the Treatment Arm and intra-aortic balloon pump (IABP) in the Control Arm).
All Stroke | At hemodynamic stability when the subject is no longer hospitalized
Minor Bleeding | At hemodynamic stability when the subject is no longer hospitalized
Minor Vascular Complications | At hemodynamic stability when the subject is no longer hospitalized
Minor Hemolysis | At hemodynamic stability when the subject is no longer hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Navin Kapur, MD, Principal Investigator — Tufts Medical Center; William O'Neill, MD, Principal Investigator — Henry Ford Health System; Gregg Stone, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (7):
- New Mexico Heart Institute, Albuquerque, New Mexico, United States
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- Germany (4):
  - Herzzentrum Dresden, Dresden, Saxony
  - University Hospital Düsseldorf, Düsseldorf
  - Universitatsklinikum Schleswig Holstein, Kiel
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
- Inselspital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Jentzer JC, Hibbert B. Optimal patient and mechanical circulatory support device selection in acute myocardial infarction cardiogenic shock. Lancet. 2024 Sep 14;404(10457):992-993. doi: 10.1016/S0140-6736(24)01588-5. Epub 2024 Sep 2. No abstract available. PMID 39236724